CLINICAL TRIAL: NCT03581747
Title: Assessment of Skin Epithelial Barrier Defects in Patients With Allergic Skin Disorders by Electrical Impedance Spectroscopy
Brief Title: Detection of Skin Epithelial Barrier in Patients With Allergic Skin Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swiss Institute of Allergy and Asthma Research (Other)
Collaborators: CK-CARE (Christine Kühne - Center for Allergy Research and Education) (Unknown); SciBase AB (Other)
Responsible Party: Sponsor
Other Study IDs: EB/EIS
Record Dates: First submitted 2018-04-25; First posted 2018-07-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-07

CONDITIONS: Atopic Dermatitis; Skin Inflammation
Keywords: Atopic dermatis; Epithelial barrier; Electrical impedance spectroscopy; Allergy
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects with atopic dermatitis
  Interventions: Device: Nevisense
- Controls
  Interventions: Device: Nevisense

INTERVENTIONS:
Device: Nevisense — Measurement of electrical impedance

SUMMARY:
The primary function of epithelial tissues is to form a barrier between the body and the external environment, in order to protect the internal tissues from environmental stresses, by minimizing water loss and preventing the entry of pathogens, pollutants and allergens. Allergic disorders, such as atopic dermatitis, have been associated to an impaired epithelial barrier function. Indeed, defects in the epithelial barriers allow tissue-damaging factors to enter the tissue and thus activate the immune response. This study aims to establish a method to assess the epithelial barrier function in vivo by electrical impedance (EI) spectroscopy, a new technique for the characterisation of epithelial tissue. By this technique, a harmless electrical signal is sent through the skin and the response of the tissue is analysed, which is influenced by several cellular properties, such as shape, orientation and size. In order to validate this technique, skin of mice was treated with some molecules able to destroy the epithelial barrier. The investigators observed that, after damaging the barrier, a decrease of the EI can be detected, consistent with the type and degree of the damage.

Based on this result, the investigators believe that this technique is a good candidate as an in vivo method to determine skin barrier defects, which might be used in the future as an early diagnostic tool for the prediction of the risk to develop atopic dermatitis in young subjects, allowing the possibility to apply in time possible preventive measures. In addition, this technique might be suitable for the evaluation of a given therapy during the hospitalisation. To confirm this hypothesis, in the present study patients with atopic dermatitis will be recruited. EI measurements will be performed in both lesional and non-lesional skin and values will be compared in order to detect any difference in the electrical response due to the inflammatory state. In addition, in order to evaluate whether these patients have an appreciable defect in their skin electrical behaviour, the investigators will compare non-lesional and lesional skin of patients with skin of healthy volunteers. Peripheral venous blood and skin biopsies will be collected, in oder to characterise several immune cell populations, to detect specific skin barrier mutations and to measure serum cytokines and immunoglobulins. These and some other parameters and will be analysed in order to identify a possible correlation with the EI.

ELIGIBILITY:
The inclusion criteria for patients in this study are as follows:

1. Age 0 - 85 years
2. Diagnosis of atopic dermatitis and/or another disease of the atopic group
3. The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated

The inclusion criteria for healthy controls in this study are as follows:

1. Age 0 - 85 years
2. No diagnosis or history of allergic disease
3. The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated Written consent will be obtained after detailed information of the study was given to the participant.

Exclusion criteria:

Unable to give consent or refusal to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Hochgebirgsklinik in Davos Wolfgang. Healthy controls will be recruited within the heathy population. All individuals will be sampled for skin, blood and other samples after informal consent.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of electrical impedance values between lesional and non-lesional skin in patients with atopic dermatitis | At Day 0 on hospital admission
  In patients with atopic dermatitis electrical impedance will be measured. Measurements will be performed in both lesional skin and non-lesional skin and values will be compared in order to detect any difference in skin permeability and electrical response due to the inflammatory state.
Comparison of electrical impedance values in healthy controls and patients with atopic dermatitis | At Day 0 on hospital admission
  In order to evaluate whether patients have an appreciable defect in their skin electrical behaviour, we will compare the skin of patients with the skin of healthy volunteers.

SECONDARY OUTCOMES:
Correlation between electrical impedance measurements and innate and adaptive immune responses | At Day 0 on hospital admission; at Day 10; at Day 20 on completion of treatment.
  50 ml of peripheral venous blood will be taken in lithium heparin 7 ml tubes and one 7 ml tube without anticoagulant for serum collection. Peripheral blood mononuclear cells (PBMC) will be purified by ficoll density gradient from venous blood and then analysed by multicolor flow cytometry, to characterize T cells, B cells, Natural Killer cells and other immune cell populations. Possible correlations between EI values and these cell subsets will be described.
Correlation between electrical impedance measurements and genes associated with epidermal barrier defects | At Day 0 on hospital admission; at Day 10; at Day 20 on completion of treatment.
  From venous blood, DNA will be isolated to detect specific skin barrier mutations, such as filaggrin defects. Possible correlations between EI values and these defects will be identified.
Correlation between electrical impedance measurements and immune biomarkers in serum | At Day 0 on hospital admission; at Day 10; at Day 20 on completion of treatment.
  From serum, cytokines and immunoglobulins will be measured, by using protein analysis methods (immunoblotting, ELISA), in order to identify a possible correlation between EI values and specific serum biomarkers.
Correlation between electrical impedance measurements and the expression profile of relevant proteins at skin tissue level | At Day 0 on hospital admission; at Day 10; at Day 20 on completion of treatment.
  Skin biopsies will be collected, Real Time Polymerase Chain Reaction (PCR) and immunohistochemistry will be performed to analyse relevant skin molecules, such epidermal barrier proteins and tight junction proteins. Possible correlations between EI values and the expression of these proteins will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Institute of Allergy and Asthma Research (SIAF), Davos Platz, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided